CLINICAL TRIAL: NCT06738576
Title: Phase II Clinical Trial to Determine the Safety and Efficacy of the Allogeneic Use of Expanded Mesenchymal Stem Cells Derived From Adipose Tissue (HC106) in the Local Treatment of Female Urinary Incontinence in Women Over 50 Years of Age
Brief Title: Allogeneic Use of Expanded Mesenchymal Stem Cells Derived From Adipose Tissue (HC106), Female Urinary Incontinence Women Over 50 Years Old
Acronym: SUITH)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUITH; 2024-514833-39-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-03; First posted 2024-12-17 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Urinary Incontinence Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- single dose of 40 million HC016 (Experimental): They will receive 1 single dose 1 dose of 40 million cells of HC016 at a concentration of 10 million cells/mL. N=40
  Interventions: Drug: allogeneic mesenchymal stem cells
- Saline solution (Placebo Comparator): They will receive a single dose of the saline solution in which the HC016 cells are conditioned, which consists of lactated ringer's, glucosaline, sodium bicarbonate and human albumin. N=20
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: allogeneic mesenchymal stem cells — Cell implantation is carried out in the following steps:
  1. - Patient anesthesia
  2. - Identification of the external urinary sphincter and the incompetent area responsible for incontinence through intraurethral cystoscopy.
  3. - Resuspension of the cells by gentle manual shaking of the vials. Once the cells are resuspended, they will be used immediately.
  4. - Injection of the cell suspension with a long, fine needle (those usually used in endoscopic puncture, <22G) at 2 points of the sphincter that will coincide with the 3 o'clock and 9 o'clock position of the hands of a clock). The injection will be superficial, trying not to go deeper than 2 mm to create a wheal in each injection visible endoscopically.
  5. - Cellular remains, if any, and the vials used will be eliminated following the usual procedures used for the management of hospital surgical waste.
  Arms: single dose of 40 million HC016
Drug: Placebo — Placebo implantation is carried out in the same way as the drug implantation
  Arms: Saline solution

SUMMARY:
Evaluate the feasibility and safety, obtaining initial efficacy data, of expanded allogeneic mesenchymal stem cells derived from adipose tissue (HC106) for the treatment of urinary incontinence in women over 50 years of age.

DETAILED DESCRIPTION:
It's a controlled trial, in phase I, proof of concept, safety and preliminary analysis of efficacy. It is planned to make 2 cohorts of patients, one with a single dose of 40 million HC016 and another group with saline solution (control).

ELIGIBILITY:
Inclusion Criteria:

* Women over 50 years old
* Women with a clinical diagnosis of genuine or mixed stress urinary incontinence (SUI) with at least 6 months of evolution. Using the definitions of urinary incontinence internationally accepted by the ICS (International Continence Society): to. SUI: any involuntary loss of urine, immediately preceded by exertion. b. Mixed UI: any involuntary loss of urine, immediately preceded by exertion or an uncontrollable desire to urinate.

The predominance of effort will be assessed when more than 50% of the patient's daily losses occur preceded by effort.

* Women in whom rehabilitative treatment has failed or patients who refuse to undergo rehabilitative or surgical treatment
* Patients without active urinary tract infection (negative urine culture) at the time of recruitment and treatment
* Signing of the informed consent form

Exclusion Criteria:

* Patients with a medical history of previous surgery for incontinence, prolapse or urological/gynecological/colorectal surgery
* Major surgery or serious trauma of the subject in the previous semester
* Women with mixed urinary incontinence, with predominant symptoms of urgency
* History of high-pressure detrusor overactivity
* Present infravesical obstruction, vesico-ureteral reflux or clinical history of urinary fistula (it will be ruled out depending on the case by urethrocystoscopy, urethrocystography and flowmetry).
* Present any malignant neoplasm, unless it is basal cell or squamous cell carcinoma of the skin, or present a history of malignant tumors, unless they have been in remission during the previous 5 years.
* Cardiopulmonary disease that, in the opinion of the investigator, is unstable or serious enough to exclude the patient from the study.
* Medical or psychiatric illness of any type that, in the opinion of the researcher, may be a reason for exclusion from the study.
* History of alcohol or other addictive substance abuse in the 6 months prior to inclusion
* Subject's allergy to anesthetics

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This trial has been designed for women, because stress urinary incontinence (SUI) predominantly affects women between 20 and 50 years of age.
Enrollment: 60 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with at least one of the complictations derived from the treatment. | 7 days
  complications derived from treatment will be considered:
  * Complications during anesthesia.
  * Complications during treatment administration.
  * Peri- and postoperative complications.
  * Adverse effects during follow-up, whether or not associated with the drug

SECONDARY OUTCOMES:
The evaluation of the PAD-test | 3 moths and 6 months
  quantification of the amount of urine lost during the duration of the test (24h),
Flowmetry values | 3 months
  improvement in the flowmetry values. It is expressed in cm3 (or ml) divided by second.and the normal values are between 50 and 80 mL/min
Quality of life SF-12 questionnaire | 3 moths and 6 months
  The score ranges between 0 and 100, where the higher score implies a better health-related quality of life Evaluate the change in the quality of life of the patients with respect to the baseline situation
Quality of life ICQ-SF questionnaire | 3 moths and 6 months
  Evaluate the change in the quality of life of the patients with respect to the baseline situation. Any score greater than zero is considered urinary incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen González Enguita, PhD, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Locations (6):
- Spain (6):
  - Hospital Universitario del Henares, Coslada, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario Doce de Octubre, Madrid, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario Infanta Elena, Valdemoro, Madrid
  - Hospital Universitario General de Villalba., Villalba, Madrid

IPD SHARING:
Plan to Share IPD: Undecided